CLINICAL TRIAL: NCT00334412
Title: AmBisome® in Combination With Caspofungin Versus AmBisome® High Dose Regimen for the Treatment of Invasive Aspergillosis in Immunocompromized Patients: Randomized Pilot Study.
Brief Title: COMBISTRAT: AmBisome® in Combination With Caspofungin for the Treatment of Invasive Aspergillosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-FR-131-0106
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — liposomal amphotericin B; Caspofungin

INTERVENTIONS:
Drug: Ambisome
Drug: caspofungin

SUMMARY:
Combination therapy of caspofungin and amphotericin B could be a useful treatment option in invasive fungal disease, but before it can be routinely recommended; carefully controlled and well-designed randomized clinical trials are needed.

DETAILED DESCRIPTION:
Efficacy and toxicity of caspofungin in combination with AmBisome® as primary or salvage treatment of invasive aspergillosis has already been assessed in patients with hematologic malignancies. Forty-eight patients with documented (n=23) or possible (n=25) Invasive Aspergillosis (IA). The majority of the patients (65%) received the combination as salvage therapy for progressive IA despite 7 or more days of previous AmBisome monotherapy. The overall response rate was 42%. No significant toxic effects were seen. Factors associated with failure at the end of therapy were documented IA (P=0.03), significant steroid use before the study (P=0.02), and duration of combination therapy for less than 14 days (P=0.01). The response rate in patients with progressive documented IA was low (18%). Authors' concluded that combination is a promising therapy for IA and was generally well tolerated.35 Furthermore interaction of caspofungin and amphotericin B for clinical isolates of Aspergillus and Fusarium was assessed. Antagonism was not observed for any of the isolates tested. Caspofungin and amphotericin B were synergistic or synergistic to additive for at least half of the isolates studied.36 Gentina et al. evaluated, in refractory IA, i.v. antifungal therapies combining caspofungin (70 mg on D1, followed by 50 mg/d) with Vfend® (200 mg b.i.d) or AmBisome (5 mg/kg/d). Six leukaemia patients with refractory IA received combination including caspofungin with AmBisome (n = 4) or Vfend (n = 2). Combination therapies were started 8 days after initial IA diagnosis. Duration of neutropenia after initiation of combination therapy ranged 4 to 25 days. IA was classified as definite in 3 cases and probable in 3 cases. All patients had pulmonary IA, including one with disseminated IA (cerebral, thyroid, ocular and pulmonary). In all patients, sequential CT-scans demonstrated improvement with a rapid reduction of the size of lesions. Additional surgery was only required in 2 cases. Improvement allowed administration of consolidation chemotherapy in 3 patients without recurrence of IA. Median duration of combination therapy was 62 days (range 42-107). No toxicity related to this combination antifungal therapy was observed.37 The combination therapy of caspofungin and amphotericin (or liposomal amphotericin) was also assessed by Aliff et al. in a retrospective evaluation of a group of 30 patients with amphotericin-resistant pulmonary aspergillosis and other invasive fungal infections. Twenty-six patients had acute leukemia. Diagnosis was based on clinical, radiographic, and when available, microbiologic data. Response to combination antifungal therapy was graded as either favorable or unfavorable. Favorable responses included improvement of both clinical and radiographic signs of fungal pneumonia. All other responses were graded as unfavorable. Based on the EORTC criteria, the IFIs were classified as proven in 6 patients, probable in 4 patients, and possible in 20 patients. The median duration and dose of amphotericin monotherapy were 12 days (range, 4-65 days) and 7.8 mg/kg (range, 4.2-66.1 mg/kg),respectively. The median duration of combination therapy was 24 days (range, 3-74 days). Eighteen patients (60%) experienced a favorable antifungal response. Twenty patients with acute leukemia received combination therapy for fungal pneumonias arising during intensive chemotherapy treatments. Favorable responses were observed in 15 of these patients (75%), and antifungal response did not depend on the response of the underlying leukemia. Survival to hospital discharge was significantly better (P < 0.001) in patients having a favorable response. Authors concluded that the combination of caspofungin and amphotericin B can be administered safely to high-risk patients with hematologic malignancies.38 Combination therapy could be a useful treatment option in invasive fungal disease, but before it can be routinely recommended; carefully controlled and well-designed randomized clinical trials are needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children > 10 years old.
* The patient is able to understand and has signed a written informed consent OR the parent or legal guardian is able to understand and has signed a written informed consent, which must be obtain prior to the initiation of any study procedures.
* Immunocompromised due to hematologic malignancies, chemotherapy-induced neutropenia, solid organ transplantation, other conditions resulting in severe neutropenia, HIV infection, prolonged corticosteroid therapy (≥ 20 mg Prednisone or equivalent for ≥ 3 weeks) or treatment with other immunosuppressant medications.
* Evidence of Proven or Probable Invasive Aspergillosis, by modified EORTC criteria (Appendix 2), as modified below: • Proven Invasive Aspergillosis • Histopathologic or cytopathologic examination showing hyphae consistent with the presence of aspergillus from needle aspiration or biopsy specimen with evidence of associated tissue damage (either microscopically or unequivocally by imaging); or • Positive culture result for aspergillosis from a sample obtained by sterile procedure from normally sterile and clinically or radiologically abnormal site consistent with infection, excluding urine and mucous membranes • Probable Invasive Aspergillosis • At least 1 host factor criterion; and • 1 microbiological criterion; and
* 1 major (or 2 minor) clinical criteria from abnormal site consistent with infection; and • No other pathogens detected to account for the clinical or radiographic signs of infection
* Or (Modification of EORTC Criteria): • Patients with recent Neutropenia (absolute neutrophil count < 500 cells/mm3 within 14 days of study enrollment); and • Chest CT scan positive for "Halo" or "Air Crescent" Sign (see Section 4.2.1, Diagnostic Considerations, below) and • No other pathogens detected to account for the clinical or radiographic signs of infection
* Females of childbearing potential must be surgically incapable of pregnancy, or practicing an acceptable method of birth control with a negative pregnancy test (blood or urine) at baseline.

Exclusion Criteria:

Life expectancy < 30 days

* Allogenic stem cell transplant in the 6 previous months
* Chronic invasive fungal infection, defined as signs/symptoms of invasive fungal infection present for > 4 weeks preceding entry into study
* Prior anti-fungal systemic therapy of ≥ 96 hours for the current, documented IA. (On the other hand, is permissible prior systemic anti-fungal therapy for prophylaxis or as empiric therapy for febrile neutropenia).
* Use of another investigational, unlicensed drug within 30 days of screening or concurrent participation in another clinical trial using an investigational, unlicensed drug • Serum creatinine > 2x upper limit of normal (ULN)
* Serum ALT or AST > 5 x ULN
* Pregnant or lactating women
* History of allergy or serious adverse reaction to any polyene anti-fungal agent or echinochandin derivatives

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-03; Study Completion 2006-05

PRIMARY OUTCOMES:
To assess efficacy of AmBisome® in combination with caspofungin (Cancidas®) versus AmBisome® high dose regimen in the treatment of Invasive Aspergillosis diagnosed by modified EORTC criteria in immunocompromised patients as probable or proven and deter

SECONDARY OUTCOMES:
To evaluate and compare the safety and tolerability of the two arms.
To determine the survival rates and rates of infection relapse at 4 weeks post-treatment for patients treated with each of the two treatment regimens.
To determine the survival rate at 12 weeks after study entry for patients treated with each of the two treatment regimens.
To determine and compare the time to favorable response and time to maximal overall response for each of the two treatment regimens.
To compare the efficacy of each arm versus historical data on conventional amphotericin B and voriconazole for the treatment of Invasive Aspergillosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lamine Mahi, MD, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Paris, France